CLINICAL TRIAL: NCT04029246
Title: Reengaging Patients With Previously Diagnosed Hepatitis C in to Care
Brief Title: Re-engaging Patients With Hepatitis C Into Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Glasgow Royal Infirmary (Other)
Collaborators: Glasgow Caledonian University (Other)
Responsible Party: Principal Investigator, stephen t barclay, Consultant Hepatologist, Glasgow Royal Infirmary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: GN19ID200
Record Dates: First submitted 2019-07-15; First posted 2019-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Letter only (No Intervention)
- Letter plus phone call (Active Comparator)
  Interventions: Behavioral: Follow up phone call
- Letter plus incentive (Active Comparator)
  Interventions: Behavioral: Incentive

INTERVENTIONS:
Behavioral: Follow up phone call — Telephone call to ask if patient has received letter and whether they would like an appointment
  Arms: Letter plus phone call
Behavioral: Incentive — Offer of a shopping voucher if patient attends for appointment
  Arms: Letter plus incentive

SUMMARY:
Aims:

To evaluate the impact of a letter, phone call and incentive in re-engaging patients with hepatitis C care.

Outcomes of interest:

Primary outcome of interest:

- Attendance for assessment of liver disease within 4 months of being sent invitation letter.

Secondary outcomes of interest:

- Commencing treatment within 6 months of being sent invitation letter.

Methods:

Patient identification:

The local copy of the Scottish Hepatitis C database holds data regarding patients referred to secondary care for treatment of their hepatitis C, and holds ethics approval for research on treatment and patient outcomes. This will be used to identify patients with hepatitis C infection that is untreated, treatment has been unsuccessful, or the patient has been treated but the outcome is unknown (due to non attendance for blood tests). The database has been cross checked with virus lab results, to ensure infection status is up to date. Finally, the patient data has been checked by NHS GG&C information team, to exclude patients who are deceased, or whom are no longer resident in NHS greater Glasgow and Clyde based on updated details obtained from SCIstore.

Inclusion criteria:

Patients (16 years and over) who have previously engaged with Hepatitis C services in Glasgow but who are either untreated, have been treated unsuccessfully, or have been treated but have not attended for blood tests to check for treatment success.

Exclusion criteria:

Patients with HIV. Patients no longer resident within NHS Greater Glasgow and Clyde area.

Allocation to contact groups:

Patients will be randomly distributed into 3 groups:

1. Letter: Will be sent letter 1 (appendix)
2. Letter plus telephone call: will be sent letter 2 (appendix) and be followed up with a telephone call from the treatment centre if no contact has been received after 4 weeks
3. Letter plus incentive: will be sent letter 3 (appendix)

Process:

Patient letters will be sent out by GG&C public health. For all 3 groups the letter will be sent with the small Hepatitis C Scotland booklet "Hepatitis C treatments have changed".

Letters will identify include the telephone number for the identified treatment centre which will be either, the last known treatment centre or a more local treatment centre were appropriate based on current residence.

Primary and secondary outcomes measures will be collected via the Scottish Hepatitis C database.

Lay Summary:

This study will test whether a letter alone, a letter plus follow up phone call or a letter with offer of incentive, will be most effective in re-engaging patients who are known to have hepatitis C but not yet received treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 years or older
* Known hepatitis C infection which is either:
* untreated
* treated but the outcome of treatment unknown

Exclusion Criteria:

* Known HIV infection
* No longer resident within NHS Greater Glasgow and Clyde area

Ages: 16 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Rate of attendance for liver assessment | 4 months
  Rates of attendance for assessment of liver disease within a 4 month period, recorded as a binary (yes/no) outcome

SECONDARY OUTCOMES:
Rates of initiation of Hepatitis C treatment | 6 months
  Rates of initiation of treatment for hepatitis C within a 6 month period, recorded as a binary (yes/no) outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen T Barclay, MBChB, Principal Investigator — NHS Greater Glasgow and Clyde
Locations (1):
- Glasgow Royal Infirmary, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-29): https://cdn.clinicaltrials.gov/large-docs/46/NCT04029246/Prot_SAP_000.pdf